CLINICAL TRIAL: NCT01426984
Title: A Double Blind Crossover Study on the Effect of Methylphenidate on Decision-making Ability of Adults With Borderline Personality Disorder (BPD) Compared to Adults With Attention Deficit Hyperactivity Disorder (ADHD) and Healthy Adults
Brief Title: A Double Blind Crossover Study on the Effect of MPH on Decision-making Ability of Adults With BPD Compared to Adults With ADHD and Healthy Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: SHA -0011-11
Record Dates: First submitted 2011-08-28; First posted 2011-09-01 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BPD adults (Experimental): adults with Borderline Personality Disorder (BPD)
  Interventions: Drug: methylphenidate

INTERVENTIONS:
Drug: methylphenidate — a capsule containing 20 mg
  Other Names: Adults with Borderline Personality Disorder

SUMMARY:
The study assesses the effect of Ritalin on working memory,attention,and decision-making measures in adults with BPD and compares it to its effect on healthy adults and adults with BPD (using data form study SHA 01-10), in a double-blind crossover design. The investigators hypothesize that Ritalin will result in better performance in all measures.

DETAILED DESCRIPTION:
Participants will be required to arrive at the cognitive laboratory in "Shalvata" for two visits: the first visit will include obtaining informed consent, screening (as detailed below), and performing a battery of computerized tasks. The second visit will include performing of the same battery of tasks, and payment.

In one of the visits, participants will receive a capsule containing Methylphenidate or placebo (MPH; Ritalin) (dosage: 10 mg in case weight<40 kg; 30 mg in case weight>90 kg; otherwise 20 mg -( The pills will be 10mg each, and the number of pills will be administered according to the dosage stated; 1-3 pills, according to weight). Prior to performing the tasks, and in the other visit they will receive a capsule containing placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults in the age of 21-50 with diagnosed with Borderline Personality Disorder (BPD)

Exclusion Criteria:

* People diagnosed with a clinical disorder other than BPD or ADD/ADHD that may impair their performance in the tasks used in the study.
* People for whom there is a contra-indication for consuming Ritalin.
* Pregnant women and nursing women; Women participants will be required to report whether they are pregnant, and in case they are, they will not participate.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Test of Variables of Attention (TOVA) score | 20 minutes
  This test, devised by Greenberg and Kindschi (1996), is one of many continuous performance tests (CPTs), rapid reaction-time tasks in which participants have to discriminate predetermined target stimuli from distracting non-targets. CPTs, and TOVA among them, are widely used both by practitioners and investigators as an objective tool for assessing ADHD and determining beneficial medical effects (Llorente et al. 2001).
  The TOVA used here is a standardized, fixed-interval (21.6 ± 1.1 min), visual CPT.
Iowa gambling task (IGT) score | 30 minutes
  a computerized version of the Iowa Gambling Task (Bechara et al. 1994), which assesses reward learning. In this task the participant is presented with four decks of cards on the computer screen. Each card yields a reward, but might also cast a loss. In each trial, the participant selects a card out of one of the four decks by clicking on it. Consequently, the card is exposed, displaying the gain and the loss for that trial. The accumulated total amount is presented at the bottom of the screen all along, and is updated after every trial. Through contingent feedback, participants are expected to learn that decks A and B yield constant large gains but also larger losses, so that their net loss across trials is 2,500 tokens, whereas decks C and D yield smaller gains but also smaller losses, leading to a net gain across trials of 2,500 tokens
Foregone Payoff Gambling Task (FPGT) score | 30 minutes
  gambling task is a version of the IGT developed for the purpose of the current study. Two differences distinguish it from the original version - a different payoff distribution as detailed in Table 3, and a feedback method called foregone payoffs: following each choice made by the participants, they get to see not only the card chosen but also the other three cards from the three decks not chosen. This provides more information, but can also cause temptation, and may distract participants from the advantageous decks (see e.g., Yechiam et al. 2005; Yechiam and Busemeyer 2006).
Spatial Working Memory (SWM) score | 10 minutes
  CANTAB task for assessing Spatial Working Memory
digit span score | 20 minutes
  Forward and Backward digit-span task (Wechsler 1981)

CONTACTS AND LOCATIONS:
Overall Officials: Hilik Levkovitz, Prof., Principal Investigator — Shalvata MHC
Locations (1):
- Shalvata Mental Health center, Hod HaSharon, Israel